CLINICAL TRIAL: NCT00903188
Title: Impact of Cyclosporine or Steroid Withdrawal at 3 Months Post Transplantation on Graft Function, Patient Survival and Cardiovascular Surrogate Markers the First 5 Years After Renal Transplantation.
Brief Title: Calcineurin Inhibitor (CNI) Versus Steroid Cessation in Renal Transplantation
Acronym: CISTCERT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Erasme University Hospital (Other); University Hospital, Ghent (Other); University of Liege (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Prof. Dr. Jean-Louis Bosmans, University Hospital Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-005844-26
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; graft function; cardiovascular events; malignancy; cyclosporin; steroids; mycophenolate; everolimus; renal biopsies; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — Cyclosporine; Mycophenolic Acid; Methylprednisolone Hemisuccinate; Methylprednisolone; Basiliximab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine (Active Comparator): Simulect + cyclosporine + Myfortic + steroid stop at 3 months
  Interventions: Drug: cyclosporine
- Everolimus (Active Comparator): Simulect + cyclosporine (decrease dose in one week at month 3 and replace by Everolimus (Certican)) + Myfortic + steroid maintenance
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: cyclosporine — Cyclosporine (Group 1):
  basiliximab dose: 1x20 mg IV on Day 0 and 1x20 mg IV on Day 4
  Cyclosporine: 8 mg/kg PO given before surgery, followed by 2x4 mg/kg/d. C-0h levels: month 1: 150-250 ng/ml; month 2: 100-200 ng/ml; month 3: withdrawal steroids: 100-150 ng/ml.
  C-2h levels: month 1: 900-1100 ng/ml; month 2: 800-1000 ng/ml; month 3: withdrawal steroids: maintain level of 750 ng/ml
  Enteric-coated mycophenolate(MPA):720mg PO pre-operatively followed by 1.44 g/day.
  Steroids: pre-operatively: 250mg methylprednisolone IV; day 1:125mg IV.
  Methylprednisolone:day 2-30:PO 12mg/d; day 31-60:tapered to 8mg/d ,day 61-90 :4mg/d; Month 3:stop
  Other Names: Neoral; Myfortic; Solumedrol; Medrol; Simulect
  Arms: Cyclosporine
Drug: Everolimus — Everolimus (Group 2):
  Basiliximab dose: idem as in group 1
  Cyclosporine: first three months idem group 1; month 3: decreased dose by 50%, simultaneously initiate everolimus at a starting dose of 0.75 mg bid.
  Once the everolimus blood levels range 6 - 12 ng/ml, cyclosporine will be stopped.
  Enteric-coated mycophenolate (MPA) dosing idem as group 1.
  Everolimus starting dose: 0.75 mg bid, trough levels: 6-12 ng/ml.
  Steroid dosing: idem group 1, but maintained at 4 mg methylprednisolone after day 60.
  Other Names: Certican; Neoral; Myfortic; Solumedrol; Medrol; Simulect
  Arms: Everolimus

SUMMARY:
This study intends to determine whether steroid withdrawal or calcineurin inhibitor withdrawal is superior for graft function and graft survival. Secondary endpoints for this study are: incidence of tumors and cardiovascular events.

The primary objective: To assess if superior graft function (glomerular filtration rate (GFR) difference of 10 ml/min) will be achieved at 1 year after transplantation in cohorts of de novo kidney transplant patients treated with Myfortic-everolimus plus steroids compared to Myfortic-cyclosporine.

DETAILED DESCRIPTION:
Methodology:

* A 5-year, multicentre, prospective, randomized, open-label, controlled study

  * Group 1: Simulect + cyclosporine + Myfortic + steroid stop at 3 months
  * Group 2: Simulect + cyclosporine (decrease dose in one week at month 3 and replace by everolimus) + Myfortic + steroid maintenance.
* In both groups MPA AUC monitoring will be done at 5-7 days and at 3 months, to ensure sufficient MPA protection.

Sample size calculations:

A total of 152 patients will be randomized (76 patients per group)

Population:

De novo kidney transplant recipients.

Study duration:

1.5 years inclusion+ follow-up during the first 5 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female recipients of a de novo kidney transplant, aged above 18 years
* Women of childbearing potential must have a negative serum or urine pregnancy test with sensitivity equal to at least 50 mIU/ml
* Patients must be capable of understanding the purpose and risks of the study, and must sign an informed consent form

Exclusion Criteria:

* Multiple organ transplantation (e.g., Kidney-pancreas, kidney-heart, kidney- liver,...)
* Transplantation of a patient who got another organ transplant previously
* Recipients of a HLA-identical living-related renal transplant
* Patients with PRA > 30%, patients who have lost a first graft from rejection within two years after transplantation, and African European patients.
* Patients with primary renal disease at risk for recurrence: FSGS, MPGN, HUS
* Pregnant or lactating women
* WBC < 2.5 x 109/l (IU), platelet count < 100 x 109/l (IU), or Hb < 6 g/dl at the time of entry into the study
* Active peptic ulcer
* Severe diarrhea or other gastrointestinal disorder, which might interfere with their ability to absorb oral medication, including diabetic patients with previously diagnosed diabetic gastroenteropathy
* Known HIV-1 or HTLV-1 positive tests
* The use of investigational drugs or other immunosuppressive drugs, as those specified in this protocol
* Patients receiving bile acid sequestrants
* Psychological illness or condition, interfering with the patient's compliance or ability to understand the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
To assess if superior graft function (GFR difference of 10 ml/min) will be achieved at 1 year after transplantation in cohorts of de novo kidney transplant patients treated with Myfortic-everolimus plus steroids compared to Myfortic-cyclosporine. | 1 year

SECONDARY OUTCOMES:
To compare the evolution of graft function (estimated GFR by means of modified MDRD formula)during the first 5 years post transplantation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Bosmans, MD/PhD, Principal Investigator — University Hospital Antwerp - Department Nephrology-Hypertension
Locations (5):
- Belgium (5):
  - Erasme University Hospital, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Antwerp, Edegem
  - University Hospital, Ghent, Ghent
  - University Hospital of Liege, Liège

REFERENCES:
- [Derived] Pipeleers L, Abramowicz D, Broeders N, Lemoine A, Peeters P, Van Laecke S, Weekers LE, Sennesael J, Wissing KM, Geers C, Bosmans JL. 5-Year outcomes of the prospective and randomized CISTCERT study comparing steroid withdrawal to replacement of cyclosporine with everolimus in de novo kidney transplant patients. Transpl Int. 2021 Feb;34(2):313-326. doi: 10.1111/tri.13798. Epub 2020 Dec 31. PMID 33277746